CLINICAL TRIAL: NCT04572035
Title: Feasibility, Acceptability and Effectiveness of a Structured Exercise + Psychoeducation Program for Students With Depression - A Proof of Concept Study
Brief Title: Exercise + Self-Compassion Intervention for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Eva Pila, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0000-E
Record Dates: First submitted 2020-09-22; First posted 2020-10-01 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise only (Experimental): Undergraduate peer-facilitators part of a curricular kinesiology program will facilitate a personalized group-based exercise program adapted to the participant's abilities, teach participants how to exercise, and gauge exercise intensity in a safe manner (26). The CANMAT guidelines will be implemented, with the program consisting of supervised group-based moderate-intensity exercise sessions lasting 30-minutes (plus 10-minutes for warm-up and cool-down), 3 times weekly, for a period of 10-weeks. Participants will start exercising at a low intensity and progressively increase until they are consistently exercising at a moderate intensity. As a result of the uncertainty surrounding the pandemic, the intervention will be conducted either via a virtual platform or in-person at the Exercise and Health Psychology Lab, depending on the health and safety restrictions applicable to when the student enrolls and begins their program.
  Interventions: Other: Exercise
- Exercise + Self-compassion (Experimental): Participants will undergo the same exercise program as described in the exercise only treatment arm. Participants will receive equal contact supplemental individual manualized strategies each session (+15-20 minutes) centered on self-compassion strategies (i.e., mindfulness, self-directed kindness meditations, and writing tasks).
  Interventions: Behavioral: Self-compassion psychoeducation; Other: Exercise
- Exercise + Behavioural Coaching (Experimental): Participants will undergo the same exercise program as described in the exercise only treatment arm. Participants will receive equal contact supplemental individual manualized strategies each session (+15-20 minutes) centered on behaviour change strategies (i.e., action planning, implementation intentions, relapse prevention, and goal setting).
  Interventions: Behavioral: Behavioural Coaching; Other: Exercise

INTERVENTIONS:
Behavioral: Behavioural Coaching — behaviour change strategies (i.e., action planning, implementation intentions, relapse prevention, and goal setting)
  Arms: Exercise + Behavioural Coaching
Behavioral: Self-compassion psychoeducation — self-compassion strategies (i.e., mindfulness, self-directed kindness meditations, and writing tasks)
  Arms: Exercise + Self-compassion
Other: Exercise — aerobic exercise program either delivered in a laboratory setting or via Zoom

SUMMARY:
An alarming number of students report depressive symptoms that make it difficult to function academically. Previous research has indicated that exercise can be effective in treating mild-moderate depression. However, individuals with depression may struggle psychologically to adhere to exercise programs. Researchers have highlighted the potential role of self-compassion, a psychological approach that is useful in dealing with personal inadequacies, to facilitate health behaviour regulation. Behavioural coaching is another approach that consists of self-regulatory strategies such as action planning and less emphasis on emotion-focused strategies. The purpose of this study is to test the effectiveness of a structured exercise and psychoeducation program on improving depressive symptoms among inactive students with depression and to evaluate if the addition of psychological components (self-compassion or behavioural coaching) affects this effectiveness. Students with mild-to-moderate depression will refer themselves to participate or be referred/recommended by Student Health Services at Western University. The study will consist of attending 3 exercise + psychoeducation sessions per week for 10-weeks. Study participants will be randomly allocated to one of three groups; exercise only, exercise + self-compassion, or exercise + behavioral coaching. All will complete questionnaires before, after, and 3-months following the end of their sessions. It is expected that participants in the exercise + self-compassion or exercise + behaviour coaching groups will show greater improvements in their depressive symptoms, program adherence and follow-up exercise behaviour and depression after 3 months than the exercise only group and that the exercise + self-compassion group will be superior to the exercise + behavioural coaching group in those measurements.

DETAILED DESCRIPTION:
This is a 10-week randomized parallel study assessing the effectiveness of exercise in reducing depressive symptoms among students with mild-to-moderate depression. This study has three treatment arms: exercise; exercise + self-compassion; exercise + behavioral coaching. Each participant will be invited to attend 3 supervised group-based sessions each week either virtually through Zoom or in-person at the Exercise and Health Psychology Lab for 10 weeks. Senior undergraduate Kinesiology students will facilitate a personalized exercise program adapted to the participant's abilities, teach participants how to exercise, and gauge exercise intensity in a safe manner. The CANMAT guidelines will be implemented, with the program consisting of supervised moderate-intensity exercise sessions lasting 30-minutes (plus 10-minutes for warm-up and cool-down), 3 times weekly, for a period of 10-weeks. Participants will start exercising at a low intensity and progressively increase until they are consistently exercising at a moderate intensity. The exercise intervention will integrate moderate intensity aerobic and resistance training activities while accounting for the physical abilities and interests of the individual participant and theh group.The exercise + psychoeducation groups will receive equal contact supplemental individual manualized strategies each session (+15-20 minutes) centered either on behaviour change strategies (i.e., action planning, implementation intentions, relapse prevention, and goal setting) or self-compassion strategies (i.e., mindfulness, self-directed kindness meditations, and writing tasks). The manualized psychoeducation sessions will be group-based with the trainer that is supervising the exercise sessions. Participants will fill out surveys before, after and three months following the intervention period.

ELIGIBILITY:
Inclusion Criteria:

Informed of the nature of the study and have agreed to and are able to read, review, and sign the informed consent form. The informed consent document will be written in English; therefore, the volunteer must have the ability to read and communicate in English.

* Student participants 17 to 30 years of age, inclusive, at the time of screening.
* Available and able to attend 3x group-based exercise training sessions per week.
* Patient Health Questionnaire (PHQ)-9 score of >5
* Godin Leisure-Time Exercise Questionnaire score of <14
* Able to engage in physical activity as assessed by the PAR-Q
* For Virtual Intervention Only: access to reliable internet connection and computer with a camera for the purpose of the Zoom Video calls

Exclusion criteria:

* Participant receives pharmacological (i.e. medications listed in list of prohibited medications document) or psychotherapy treatment for depression or anxiety
* Reports of suicide ideation (e.g., PHQ-9 item) and scores on the PHQ-9 >20 demonstrating severe depression
* Failed safety screening for exercise without physician clearance
* Participant initiates pharmacological or psychotherapy treatments for depression while in the study and/or participates in any other research that aims to target depression

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention (recruitment) | From recruitment to baseline
  Proportion of screened individuals choosing to participate (and reasons for not participating)
Feasibility of intervention (compliance) | From baseline to 3-month follow-up
  Proportion of program sessions attended (and reasons for non-attendance); proportion of participants that complete surveys
Feasibility of intervention (completion) | From baseline to 3-month follow-up
  Proportion of participants who drop-out prior to program completion
Feasibility of intervention (delivery) | From recruitment to post-intervention
  Proportion of eligible peer facilitators that maintain their participation in the full intervention
Acceptability of intervention | Post-intervention
  Treatment Acceptability Questionnaire - mean score ranging from 1 (low acceptability) to 7 (high acceptability)
Effectiveness of intervention (depressive symptoms) | From baseline to 3-month follow-up.
  Change in depressive symptoms measured by Patient Health Questionnaire 9 - total score ranges from 0 (no symptoms) to 27 (severe symptoms) for all treatment arms
Effectiveness of intervention (exercise behaviour) | From baseline to 3-month follow-up.
  Change in exercise measured by Leisure Time Exercise Questionnaire - calculate Leisure Score Index with higher values indicating higher exercise frequency/intensity for all treatment arms

SECONDARY OUTCOMES:
Effectiveness of psychological component (depressive symptoms) | From baseline to 3-month follow-up.
  Treatment arm difference in changes in depressive symptoms measured by Patient Health Questionnaire 9 - total score ranges from 0 (no symptoms) to 27 (severe symptoms)
Effectiveness of psychological component (exercise behaviour) | From baseline to 3-month follow-up.
  Treatment arm difference in changes in exercise behaviour measured by Leisure Time Exercise Questionnaire - calculate Leisure Score Index with higher values indicating higher exercise frequency/intensity
Effectiveness of psychological component (compliance) | From baseline to 3-month follow-up.
  Treatment arm difference in compliance (attendance in program sessions)

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] KARVONEN MJ, KENTALA E, MUSTALA O. The effects of training on heart rate; a longitudinal study. Ann Med Exp Biol Fenn. 1957;35(3):307-15. No abstract available. PMID 13470504
- [Background] Prapavessis H, De Jesus S, Fitzgeorge L, Faulkner G, Maddison R, Batten S. Exercise to Enhance Smoking Cessation: the Getting Physical on Cigarette Randomized Control Trial. Ann Behav Med. 2016 Jun;50(3):358-69. doi: 10.1007/s12160-015-9761-9. PMID 26791022
- [Background] Ravindran AV, Lam RW, Filteau MJ, Lesperance F, Kennedy SH, Parikh SV, Patten SB; Canadian Network for Mood and Anxiety Treatments (CANMAT). Canadian Network for Mood and Anxiety Treatments (CANMAT) Clinical guidelines for the management of major depressive disorder in adults. V. Complementary and alternative medicine treatments. J Affect Disord. 2009 Oct;117 Suppl 1:S54-64. doi: 10.1016/j.jad.2009.06.040. Epub 2009 Aug 8. PMID 19666194